CLINICAL TRIAL: NCT03090763
Title: Role of Circulating MicroRNAs in Pathogenesis of Aneurysms of the Abdominal and Thoracic Aorta - Study "Micro AAA"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Ass. prof. Jean-Claude M. Lubanda, MD, Ph.D, Ass.prof., Charles University, Czech Republic
Other Study IDs: Micro AAA
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Polymerase Chain Reaction; Base Sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study population: 100 Subjects followed in our department for the diagnosis of aortic aneurysm. On admission, the demographic data (see Appendix 1) will be recorded. Furthermore, within the routine clinically indicated laboratory samples, the levels of selected biochemical markers will be recorded (see Appendix 1). Follow up control laboratory will be performed one year, again within the routine samples.
  Interventions: Genetic: PCR and sequencing
- Control population: The control population also includes 100 subjects in total. These will be chosen from aged and sex matched individuals seen in our clinic without disease of the aorta. All subjects included in trial must be at least 18 years old and must sign the informed consent to participation in the study. In the control population, also demographic data will be obtained and the levels of selected biochemical markers will be recorded within the routine clinically indicated laboratory samples.
  Interventions: Genetic: PCR and sequencing

INTERVENTIONS:
Genetic: PCR and sequencing — Blood will be subsequently added into a test tube containing RNA solution of a stabilizer, necessary for preservation of the circulating miRNAs. Subsequently, centrifugation will be performed in a cooled centrifuge and the material thus processed will be kept for the subsequent isolation. The isolation of miRNA will be performed using the High Pure miRNA Isolation Kit (Roche, Basel, CHE) according to the manufacturer's standardized procedure. Presence and quality of the miRNA isolated will be spectrophotometrically confirmed using the NanoDrop device (ThermoScientific, Wilmington, DE, USA). By means of the data available in the on-line gene data basis, primers that are necessary for amplification of miRNA through the RT-PCR method using fluorescent dyes will be suggested.

SUMMARY:
The objective of this study is to establish whether patients with aortic aneurysm, compared to general population, have higher levels of selected miRNAs and whether there is significant association between the level of miRNA in circulating blood and the size of the aortic aneurysm or the risk of its rupture.

DETAILED DESCRIPTION:
Aneurysm of the abdominal and thoracic aorta represents a major cause of cardiovascular morbidity and mortality. The course of this condition can stay asymptomatic for long, and its first manifestation can be acute rupture of the aneurysm sac with life-threatening bleeding. Detection of patients at risk and their early treatment significantly reduce the percentage of this potentially lethal complications.

Aortic diseases are most often degenerative processes with a varying involvement of genetic predisposition. In literature, a substantial number of genes were proved to affect the metabolism of the vessel wall and to determine production of structural proteins, which were associated with the vascular pathologies. Pathophysiologic mechanisms of lesions of the aortic wall have not been completely understood. Among other, they include endothelial dysfunction, chronic inflammation of the vessel wall, apoptosis of smooth muscle cells and degradation of the extracellular matrix, resulting in the loss of integrity of layers of the vessel wall and decrease in its strength, which leads to dilation, rupture or dissection. Apart from mutations in genes coding the structural proteins of the vessel wall, many other potential biomarkers were proposed for early diagnosis of aortic aneurysm. These include microRNA (miRNA), one-fibre chains of non-coding ribonucleic acid which are several nucleotides long and are involved in the gene expression through the mechanism of inhibition of mRNA translation or increase in its degradation. Recently, association of levels of these miRNAs to presence and growth of aortic aneurysms has been described.

ELIGIBILITY:
Inclusion Criteria:

study population:

* signed informed consent for participation to the study;
* age above 18 years;
* presence of untreated thoracic or abdominal aortic aneurysm (TAA or AAA);
* CT-verified diagnosis of AAA/TAA including measurement of the maximum diameter of the aneurysm.

control population:

* signed informed consent for participation in the study;
* age above 18 years;
* absence of a thoracic or abdominal aortic aneurysm (TAA or AAA).

Exclusion Criteria:

* life expectation above one year;
* history of myocardial infarction or unstable angina pectoris 1 month ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * signed informed consent for participation to the study;
  * age above 18 years;
  * presence of untreated thoracic or abdominal aortic aneurysm (TAA or AAA);
  * CT-verified diagnosis of AAA/TAA including measurement of the maximum diameter of the aneurysm.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Difference in levels of circulating miRNAs | March 2017
  Difference in levels of circulating miRNAs (in ng/μl) in the population of patients with AAA/TAA compared to the control population without the aortic disease.
Correlation between the level of the circulating miRNAs and the maximal diameter of the aneurysm sac. | March 2017
  Correlation between the level of the circulating miRNAs and the maximal diameter of the aneurysm sac.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles University in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No